CLINICAL TRIAL: NCT01899885
Title: Acute High-risk Abdominal Surgery Study - an Optimized Perioperative Course
Acronym: AHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Line Toft Tengberg, MD, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHA-37855
Record Dates: First submitted 2013-07-04; First posted 2013-07-16 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Perforated Viscus; Intestinal Obstruction
Keywords: Emergency laparotomy; Emergency laparoscopy
MeSH Terms: conditions — Intestinal Obstruction | interventions — acetohydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- historic control group (No Intervention): Standard treatment in the historic control group
- Intervention group (Active Comparator): AHA (Acute Highrisk Abdominalsurgery): Optimized Course:
  Intervention before, during and after abdominal surgery.
  Focus on fast track with multimodal standardized intervention:
  1. standardized preparing for surgery including high dose antibiotics and epidural analgesia etc. and transfer to intermediate care before surgery (the post-anaesthesia care unit)
  2. GDT-LiDCO fluid management pre-, per- and postoperative
  3. Postoperative triage to 24 hour intermediate care based on ASA score and Surgical Apgar Score
  4. Focus on early mobilization, fysiotherapy and optimal nutrition postoperatively
  Interventions: Procedure: AHA (Acute Highrisk Abdominalsurgery): Optimized Course

INTERVENTIONS:
Procedure: AHA (Acute Highrisk Abdominalsurgery): Optimized Course — optimized course: Intervention before, during and after abdominal surgery.
  Focus on fast track with multimodal standardized intervention:
  1. standardized preparing for surgery including high dose antibiotics and epidural analgesia etc. and transfer to intermediate care before surgery (the post-anaesthesia care unit)
  2. GDT-LiDCO fluid management pre-, per- and postoperative
  3. Postoperative triage to 24 hour intermediate care based on ASA score and Surgical Apgar Score
  4. Focus on early mobilization, fysiotherapy and optimal nutrition postoperatively
  Arms: Intervention group

SUMMARY:
The objective of this study is to implement an optimized perioperative course for patients undergoing acute high-risk abdominal surgery in order to improve the outcome.

The optimized perioperative course consists of a number of interventions carried out before, during and after surgery.

DETAILED DESCRIPTION:
Emergency surgery is associated with high mortality rates, post-operative complications and prolonged duration of hospital admission. The investigators will implement a multidisciplinary optimized perioperative course consisting of a number of interventions carried out before, during and after surgery.

Hypothesis: An optimized perioperative course will reduce the 30-day mortality in emergency abdominal surgery patients.

The investigators will do a post-hoc analysis of the data registered.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary emergency laparotomy or laparoscopy
* patients undergoing reoperation after abdominal surgery.
* Age > 18 years

Exclusion Criteria:

* Appendectomy
* Emergency laparoscopic cholecystectomy
* Emergency diagnostic laparoscopy without intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
mortality rate | Within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Line T Tengberg, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Tengberg LT, Bay-Nielsen M, Bisgaard T, Cihoric M, Lauritsen ML, Foss NB; AHA study group. Multidisciplinary perioperative protocol in patients undergoing acute high-risk abdominal surgery. Br J Surg. 2017 Mar;104(4):463-471. doi: 10.1002/bjs.10427. Epub 2017 Jan 23. PMID 28112798